CLINICAL TRIAL: NCT05080036
Title: Muscle Activation of the Lower Limb in Healthy Subjects in Response to a Medio-lateral Imbalance in Monopodal Stance: a Preliminary Study
Brief Title: Muscle Activation of the Lower Limb in Response to a Medio-lateral Imbalance in Monopodal Stance
Acronym: SM01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manusapiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 957/2020/SPER/AUSLRE
Record Dates: First submitted 2021-08-26; First posted 2021-10-15 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: human balance; monopodal stance; electromyography; myofascial chains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unbalanced healthy subjects (Experimental): Subjects undergo an external perturbation of their balance
  Interventions: Other: Medio-lateral imbalance

INTERVENTIONS:
Other: Medio-lateral imbalance — Thrust on the pelvis in the medio-lateral direction in order to create a balance perturbation

SUMMARY:
The "static" single-leg stance has been extensively studied in the literature for its relevance in functional evaluation, therapeutic exercise, sports training and research for fall prevention (particularly for the elderly and patients with neurological diseases). However, the motor strategies of the supporting limb have been investigated only at the ankle level. In particular it is not known, at the hip, how the muscular system reacts to medial and lateral imbalances. Colonna has hypothesized, basing on a myofascial chains approach, that the balance is managed by the front and back spiral chains. The aim of the present study is to perform a preliminary experimental analysis to verify Colonna's hypothesis, testing a method for the investigation of motor strategies underlying equilibrium.

Five healthy subjects will be examined by means of electromyographic analysis of the gluteus maximus, gluteus medius, adductor longus, tibialis anterior and peroneus longus. Subjects will undergo perturbations of their monopodal balance.

DETAILED DESCRIPTION:
The subjects involved in the research will be analyzed at the LAMBDA laboratory (UDGEE), AUSL-IRCCS (Azienda Unità Sanitaria Locale-Istituto di Ricovero e Cura a Carattere Scientifico) di Reggio Emilia.

The analysis will be carried out on the right lower limb of each subject. The electromyographic devices will be applied to the tibialis anterior, peroneus longus, gluteus medius, gluteus maximus and adductor longus.

Reflective markers will then be applied (using double-sided tape) according to the Total3DGait protocol, which identifies the body segments of the forearms, arms, trunk, pelvis, thighs, legs, and feet.

The subject must position himself with his right foot on a force platform. The toe of the left foot will be allowed to rest on the ground (on the other power platform posteriorly placed), with the verbal indication to load as little weight as possible on it: this indication is aimed at reducing muscle activation in the absence of external perturbations, in order to highlight only the activity caused by the perturbations themselves. Only acquisitions in which the load on the left foot will be less than 30% of the weight will be considered valid.

The hands will be placed on the hips to limit the variables to be controlled and to standardize the posture, in order to focus the contribution to the balance of the lower limb. The left thigh has to be kept vertical. Finally, it will be required to find, within the constraints described above, the posture that is as comfortable as possible, with minimal muscle contraction. The distance between the feet is therefore freely chosen by each subject.

The operator positions himself behind the subject to be examined, and without being seen performs lateral thrusts with the medial margin of the hand at the proximal third of the thigh. At least ten pushes per side will be performed, with random timing. The thrusts will be quick but without causing pain.

The operator will then request maximal contractions from the subject, in order to normalize the electrical activity of each muscle with respect to its maximum. It will be required to perform the dorsiflexion and pronation of the foot against resistance, then the adduction, abduction and extension of the hip.

ELIGIBILITY:
Inclusion Criteria:

* All healthy subjects

Exclusion Criteria:

* skeletal pathologies compromising balance
* neuromotor pathologies compromising balance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum electrical intensity during early response of muscle activation | During the procedure
  The muscles considered will be, for the anterior spiral chain, the adductor longus and the peroneus longus, for the posterior spiral chain, the glutei (medius and maximus) and the tibialis anterior. For each muscle, the intensity will be normalized to the intensity of the maximal contraction. Muscle activity will be evaluated for 1500ms, 500ms before and 1000ms after the thrust. The early response to the stimulus will be identified in the interval of 100-500ms after the thrust.The thrusts will be performed 10 times towards the medial direction and 10 towards the lateral. The median intensity for each direction will be calculated.
Correlation of muscle activity | During the procedure
  Correlation coefficients of the activation intensity between each muscle of the hip and each muscle of the ankle: tibialis anterior-glutei; tibialis anterior-adductor longus; peroneus longus-glutei; peroneus longus-adductor longus. Calculated for each imbalance direction.

CONTACTS AND LOCATIONS:
Locations (1):
- AUSL-IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colonna S., 2012. Le catene miofasciali in medicina manuale - Arto inferiore: Ginocchio, Ed. Martina.
- [Background] Morey-Klapsing G, Arampatzis A, Bruggemann GP. Joint stabilising response to lateral and medial tilts. Clin Biomech (Bristol). 2005 Jun;20(5):517-25. doi: 10.1016/j.clinbiomech.2005.01.008. PMID 15836939

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT05080036/Prot_SAP_000.pdf